CLINICAL TRIAL: NCT00823030
Title: Effect of Intravesical Lidocaine on Urodynamic and Symptomatic Parameters of Interstitial Cystitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Robert Moldwin, principal investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 08-221
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Interstitial Cystitis
Keywords: Interstitial Cystitis; Intravesical Lidocaine
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo instillation: 20 ml of normal saline instilled intravesically
  Interventions: Procedure: Urodynamic study; Other: Normal Saline
- experimental arm (Experimental): The experimental instillation will include 8 ml of 2% lidocaine, 3 ml of sodium bicarbonate, and 9 ml of normal saline.
  Interventions: Procedure: Urodynamic study; Drug: Lidocaine

INTERVENTIONS:
Procedure: Urodynamic study — A small catheter will be inserted into the bladder and water will slowly be instilled through the catheter and into your bladder. A series of measurements will then be taken to assess your bladder's capacity to hold liquid, the average and maximum urine flow rates, as well as bladder filling and leak point pressure readings.
  Other Names: UDS
Drug: Lidocaine — 20 cc of alkalinized lidocaine will be injected after the first UDS
  Arms: experimental arm
Other: Normal Saline — 20 cc of normal saline will be injected into the bladder after the first UDS
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the amount of improvement in bladder function and pain relief with the administration of 2% alkalinized lidocaine in patients with interstitial cystitis. Specifically, we want to see if the administration of 2% alkalinized lidocaine treatments in the bladder improves urodynamic test result values. We hope to enroll approximately 40 patients in this study.

Previous research has shown that the administration of 2% alkalinized lidocaine in the bladder may improve the bladder's capacity to hold urine and urine flow rates while simultaneously providing pain relief. As part of standard of care at the Smith Institute of Urology Pelvic Pain Center, we routinely offer our IC patients 2% alkalinized lidocaine with follow up urodynamic evaluation. Our research looks to expand upon the prior studies and confirm the findings of improved bladder function and enhanced pain control of 2% alkalinized lidocaine versus placebo by performing a second urodynamic evaluation, which is not routinely performed.

DETAILED DESCRIPTION:
Interstitial cystitis (IC) is a chronic bladder condition that includes symptoms of bladder or pelvic pain as well as irritative voiding symptoms (urgency, frequency, nocturia, dysuria). The syndrome is usually diagnosed clinically after ruling out any possible infectious or neoplastic causes. Due to the lack of standardized diagnostic criteria, the reported prevalence of IC in the United States varies widely from 35 to 24,000 per 100,000 persons1,2. Regardless, there is no doubt that IC is a source of much distress and profoundly affects quality of life. IC patients have been reported to have lower quality of life than dialysis patients. They are 6 times more likely than the general population to cut down on work time owing to health problems and have higher reported incidences of depression, chronic pain, anxiety and overall mental health2,

The exact pathophysiology or etiology of IC is not completely understood but there have been much advancement in knowledge. The etiology is most likely multifactorial and studies have shown a role for epithelial dysfunction, inflammatory events as well as neurological dysfunction [Figure 1]. An initiating event such as infection, trauma, or autoimmune disorder leads to dysfunctional urothelium4. Activation and upregulation of sensory nerves occurs, leading to mast cell activation and release of histamine and other mediators5,6. This, in turn, leads to a cycle of symptoms for the IC patient.

Due to the multifactorial nature of its pathogenesis, IC treatment is complicated and involves multimodal treatments that target different factors. Tricyclic antidepressants control the regulation and activation of the nerves7. Antihistamines target mast cell activation8 while heparinoids such as pentosan polysulfate sodium (PPS) or heparin targets the dysfunction epithelium. Heparin is one of the most commonly used intravesical agent for the treatment of IC. It has been found to be effective is almost 50% of patients9. While heparinoid therapy enhances the barrier effect of the disrupted urothelium, it does not directly target the sensory nerves of the bladder. Hence, it may take more than 2 years of treatment for severely affected patients to feel any symptomatic relief10. Furthermore, once symptomatic relief is achieved, it is not sustained for very long11. Urologists aimed to develop therapy that would directly affect the sensory nerves of the bladder and provide immediate symptomatic relief.

The use of intravesical lidocaine in severe IC was first reported in Sweden in 1989. Asklin et al., reported on one patient who received repeated intravesical instillations of lidocaine and achieved much relief13. Success with the treatment was subsequently reported for another patient in 199214. Surprisingly, there have been very few studies on the clinical efficacy of intravesical lidocaine in IC patients since then. To date, all studies involving intravesical lidocaine lack randomization or a control group. It is difficult to determine the influence of any existing placebo effect of intravesical instillations.

One such study was conducted in 2005 by Parsons et al., which tested the efficacy of heparin combined with intravesical lidocaine in 47 newly diagnosed IC patients. 75% of patients reported significant improvement in symptoms after just one instillation with symptomatic relief lasting at least 4 hours. Significant improvement in symptoms was reported in 94% of patients who received a second instillation using a higher concentration of lidocaine. Of 20 patients who received a course of 6 instillations over 2 weeks, 80% reported sustained relief15.

Welk and Telchman looked specifically at dyspareunia response to intravesical lidocaine in 23 IC patients. 57% reported resolution of dyspareunia. They also found a significant difference in response rate between patients with bladder tenderness and patients with multiple tender locations on vaginal exam (85% versus 29% respectively)16.

Urodynamic studies performed in IC patients generally demonstrate normal cystometry, although IC patients have characteristic reductions in bladder capacity secondary to pain and hypersensitivity to bladder dilation3. In a recent retrospective study, Srinivasan et al observed that a statistically significant difference was appreciable when comparing pre and post lidocaine UDS evaluation in bladder capacity, maximum flow rate, and first strong sensation to void. 12 The impact of alkalinized lidocaine on UDS parameters, however, remains elusive and deserving of a well designed randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18
* Clinical diagnosis of Interstitial cystitis based on the National Institute of Diabetes, Digestive and Kidney Diseases (NIDKK) criteria. According the NDIKK criteria, IC patients must have either glomerulations on cystoscopic examination or classic Hunner Ulcers and must also have either pain associated with the bladder or urinary urgency. Symptoms of abnormal urinary frequency and bladder pain/discomfort must have been present for at least 3 months prior to study entry
* Able to understand and complete a VAS/GRA/modified IPSS assessment
* Written informed consent

Exclusion Criteria:

* Currently asymptomatic
* Severely debilitating or urgent concurrent medical condition
* History of pelvic radiation therapy, tuberculous cystitis, neurologic disease affecting bladder function, bladder cancer, or carcinoma in situ, or urethral cancer
* Presence of bladder, urethral, or ureteral calculi
* Clinical evidence of urethritis
* Unlikely to be compliant due to unmanaged medical or psychological problem, including neurological, psychological or speech/language problems that will interfere with ability to complete the study
* Allergy to lidocaine or any of the other anesthetics in the amide family.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Urodynamic parameters | 2 hours, 1 baseline UDS will be checked and then another will be checked one hour after the interventional step

SECONDARY OUTCOMES:
symptom scores (Global response assessment, IPSS, VAS) | baseline, after 2nd UDS, and at 3 and 7 days after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Moldwin, M.D., Principal Investigator — Northwell Health
Locations (1):
- Smith Institute for Urology, Lake Success, New York, United States

REFERENCES:
- [Background] Parsons CL, Tatsis V. Prevalence of interstitial cystitis in young women. Urology. 2004 Nov;64(5):866-70. doi: 10.1016/j.urology.2004.06.044. PMID 15533465
- [Background] Parsons CL, Housley T, Schmidt JD, Lebow D. Treatment of interstitial cystitis with intravesical heparin. Br J Urol. 1994 May;73(5):504-7. doi: 10.1111/j.1464-410x.1994.tb07634.x. PMID 8012771
- [Background] Welk BK, Teichman JM. Dyspareunia response in patients with interstitial cystitis treated with intravesical lidocaine, bicarbonate, and heparin. Urology. 2008 Jan;71(1):67-70. doi: 10.1016/j.urology.2007.09.067. PMID 18242367
- [Background] Asklin B, Cassuto J. Intravesical lidocaine in severe interstitial cystitis. Case report. Scand J Urol Nephrol. 1989;23(4):311-2. doi: 10.3109/00365598909180345. PMID 2595329
- [Background] Parsons CL. Successful downregulation of bladder sensory nerves with combination of heparin and alkalinized lidocaine in patients with interstitial cystitis. Urology. 2005 Jan;65(1):45-8. doi: 10.1016/j.urology.2004.08.056. PMID 15667861
- [Background] Srinivasan A, Shapiro E and Moldwin RM: Effects of Intravesical Lidocaine on Urodynamic Parameters in Patients with Interstitial Cystitis/Painful Bladder Syndrome (IC/PBS).